CLINICAL TRIAL: NCT05175599
Title: Hospital Waterbirth: A Pilot Randomized Control Study
Brief Title: Hospital Waterbirth Trial to Measure Maternal and Neonatal Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00106915; 20.176 (Other: Advocate Aurora Health Care)
Record Dates: First submitted 2021-09-20; First posted 2022-01-04 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Natural Childbirth

STUDY DESIGN:
Intervention Model Description: Women are randomized 1:2 land birth to waterbirth.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Land Birth (No Intervention): Women in the land birth group will labor and give birth according to standard of care procedures.
- Water Birth (Experimental): Women in the water birth group will give birth in the water. During the first stage of labor, women may enter or leave the water at any point.
  Interventions: Other: Water Birth

INTERVENTIONS:
Other: Water Birth — The water birth group will use a tub of a water to labor and give birth.
  Arms: Water Birth

SUMMARY:
This study aims to explore outcomes of waterbirth in comparison to conventional land birth for low-risk healthy women and neonates in a hospital setting in Milwaukee, WI. This study hypothesizes that women who labor and birth in water will use less pain medication, have a shorter labor, will be more likely to initiate breastfeeding prior to discharge, will not experience more negative outcomes, and will experience greater satisfaction than women who labor and birth on land.

DETAILED DESCRIPTION:
Women eligible for a waterbirth will be randomized (2:1) to either waterbirth or land birth at the beginning of the third trimester (25 weeks 0 days to 34 weeks 0 days gestation). The investigators recognize that some women will risk-out or opt-out because of the unpredictability of labor and birth. The goal is that approximately 50% of enrolled waterbirth participants give birth in water. Additionally, the investigators aim to approach the majority of patients eligible for waterbirth with the understanding that some women will not want to participate in a research study. Please note that given the variable nature of birth, once a woman is randomized and enrolled to either group, an intention to treat model will be used for analysis. Following birth, women will be asked to complete a validated questionnaire to evaluate maternal satisfaction prior to discharge. Other data will be collected from our electronic medical record or 4-8 weeks postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Prenatal low-risk, healthy, adult women (greater than or equal to 18 years of age), including:

  1. Able to speak and understand English
  2. Women with a singleton gestation
  3. Able to ambulate with no mobility restrictions (i.e., no difficulty getting from seated to standing)
  4. Less than class III obesity (BMI <40kg/m squared) at initiation of prenatal care
  5. No active infections such as HIV, Hepatitis B, Hepatitis C, HSV outbreak (on prophylaxis acceptable), GBS positive is acceptable
  6. No pre-existing medical conditions such as: heart disease, uncontrolled asthma, diabetes of any type, chronic hypertension, or other condition that requires continuous observation and/or activity restrictions
  7. No high-risk pregnancy conditions: including preeclampsia, gestational hypertension, preterm gestation, multiple gestation, substance abuse, placental abruption or other unexplained vaginal bleeding, previous cesarean section, suspected fetal macrosomia (>4500gm) or intrauterine growth restrictions (<10th percentile), or other condition that requires continuous observation and/or activity restrictions

     Labor inclusion criteria:
  8. Greater than 37 weeks and less than 42 completed weeks gestation in vertex presentation
  9. Not hypertensive or febrile (two blood pressures 140/90 four hours apart; two fevers of over 100.4 one hour apart)
  10. Category 1 fetal heart tones (obtained on a 20-minute admission external fetal monitor strip)
  11. Amniotic sac may be intact or ruptured. If ruptured, amniotic fluid must be clear.

Exclusion Criteria:

* Women will be excluded from the study if they do not meet above inclusion criteria or they will be further excluded under the following circumstances:

  1. Known need for cesarean section
  2. Participant may be excluded from the study at any time at the discretion of the birth attendant (reason for study exclusion will be documented but will remain in the study group previously selected based on intention to treat).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

PRIMARY OUTCOMES:
Pain Medication | Time of admission to birth of the baby
  The percent of women in the waterbirth cohort who use IV narcotic and epidural anesthesia will be reduced when compared with the land birth cohort.

SECONDARY OUTCOMES:
Labor duration | Time of labor onset to time of birth
  The percent of women in the waterbirth cohort will have shorter labor duration than women in the land birth cohort.
Rate of breastfeeding | Measured from birth (immediate) through discharge from hospital (24-48 hours)
  The percent of women in the waterbirth cohort who initiate immediately after the birth breastfeeding will be higher than women in the land birth cohort.
Patient satisfaction based on the United States Birth Satisfaction Scale-Revised (US-BSS-R) | During postpartum hospital stay, starting at the time of birth until up to 72 hours from the time of birth
  Women in the waterbirth cohort will have higher scores on the US-BSS-R scale during their postpartum hospital stay (up to 72 hours after the time of birth) than women in the land birth cohort. The US-BSS-R is a 10 question scale using a 5 point Likert scale with answers ranging from "strongly agree" to "strongly disagree"
Reported maternal adverse outcomes | During labor and birth through the immediate postpartum hospital admission (24-48 hours after the birth)
  The percent of women in the waterbirth cohort with reported adverse obstetric outcomes will be less than women in the land birth cohort.
Reported neonatal adverse outcomes | Immediately after the birth until the time of the postpartum visit (usually 4 to 6 weeks of life)
  The percent of neonates in the waterbirth cohort with reported adverse birth outcomes will be less than neonates in the land birth cohort.
Instrumental and cesarean deliveries | Time of labor to time of delivery
  The percent of neonates in the waterbirth cohort with instrumental and cesarean deliveries will be less than neonates in the land birth cohort.
Skin-to-skin contact | Measured from time of birth (hour/minute) to time of skin-to-skin contact initiation (in number of minutes) up to 60 minutes of life.
  Neonates in the waterbirth cohort will have longer duration in minutes of skin-to-skin contact (on the maternal abdomen or chest) when compared with neonates in the land birth cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Malloy, CNM, APNP, Principal Investigator — emily.malloy@aah.org
Locations (1):
- Aurora Sinai Medical Center, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nutter E, Meyer S, Shaw-Battista J, Marowitz A. Waterbirth: an integrative analysis of peer-reviewed literature. J Midwifery Womens Health. 2014 May-Jun;59(3):286-319. doi: 10.1111/jmwh.12194. PMID 24850284
- [Background] Duffin C. Waterbirth findings reveal high levels of satisfaction: Royal College of Midwives annual conference reflects a further move away from medical interventions towards. Nursing Standard. 2004 May 26;18(37):8-9.
- [Background] Cluett ER, Burns E. Immersion in water in labour and birth. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD000111. doi: 10.1002/14651858.CD000111.pub3. PMID 19370552
- [Background] Cluett ER, Burns E, Cuthbert A. Immersion in water during labour and birth. Cochrane Database Syst Rev. 2018 May 16;5(5):CD000111. doi: 10.1002/14651858.CD000111.pub4. PMID 29768662
- [Background] Lawrence A, Lewis L, Hofmeyr GJ, Dowswell T, Styles C. Maternal positions and mobility during first stage labour. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003934. doi: 10.1002/14651858.CD003934.pub2. PMID 19370591
- [Background] Shaw-Battista J. Systematic Review of Hydrotherapy Research: Does a Warm Bath in Labor Promote Normal Physiologic Childbirth? J Perinat Neonatal Nurs. 2017 Oct/Dec;31(4):303-316. doi: 10.1097/JPN.0000000000000260. PMID 28520654
- [Background] ACNM. Position statement: Hydrotherapy during labor and birth. 2014.
- [Background] Committee Opinion No. 679: Immersion in Water During Labor and Delivery. Obstet Gynecol. 2016 Nov;128(5):e231-e236. doi: 10.1097/AOG.0000000000001771. PMID 27776074
- [Background] Maude RM, Foureur MJ. It's beyond water: stories of women's experience of using water for labour and birth. Women Birth. 2007 Mar;20(1):17-24. doi: 10.1016/j.wombi.2006.10.005. Epub 2006 Dec 14. PMID 17174165
- [Background] ACOG Committee Opinion No. 766: Approaches to Limit Intervention During Labor and Birth. Obstet Gynecol. 2019 Feb;133(2):e164-e173. doi: 10.1097/AOG.0000000000003074. PMID 30575638
- [Background] Dahlen HG, Dowling H, Tracy M, Schmied V, Tracy S. Maternal and perinatal outcomes amongst low risk women giving birth in water compared to six birth positions on land. A descriptive cross sectional study in a birth centre over 12 years. Midwifery. 2013 Jul;29(7):759-64. doi: 10.1016/j.midw.2012.07.002. Epub 2012 Aug 11. PMID 22884894
- [Background] Pagano E, De Rota B, Ferrando A, Petrinco M, Merletti F, Gregori D. An economic evaluation of water birth: the cost-effectiveness of mother well-being. J Eval Clin Pract. 2010 Oct;16(5):916-9. doi: 10.1111/j.1365-2753.2009.01220.x. PMID 20590979
- [Background] Odent M. Birth under water. Lancet. 1983 Dec 24-31;2(8365-66):1476-7. doi: 10.1016/s0140-6736(83)90816-4. No abstract available. PMID 6140561
- [Background] Henderson J, Burns EE, Regalia AL, Casarico G, Boulton MG, Smith LA. Labouring women who used a birthing pool in obstetric units in Italy: prospective observational study. BMC Pregnancy Childbirth. 2014 Jan 14;14:17. doi: 10.1186/1471-2393-14-17. PMID 24423216
- [Background] Chaichian S, Akhlaghi A, Rousta F, Safavi M. Experience of water birth delivery in Iran. Arch Iran Med. 2009 Sep;12(5):468-71. PMID 19722768
- [Background] Gayiti MR, Li XY, Zulifeiya AK, Huan Y, Zhao TN. Comparison of the effects of water and traditional delivery on birthing women and newborns. Eur Rev Med Pharmacol Sci. 2015;19(9):1554-8. PMID 26004591
- [Background] Woodward J, Kelly SM. A pilot study for a randomised controlled trial of waterbirth versus land birth. BJOG. 2004 Jun;111(6):537-45. doi: 10.1111/j.1471-0528.2004.00132.x. PMID 15198780
- [Background] Torkamani SA, Kangani F, Janani F. The effects of delivery in water on duration of delivery and pain compared with normal delivery. Pak J Med Sci. 2010; 26(3):551-5.
- [Background] Ghasemi, M, Tara, F., Ashraf, H. Maternal-Fetal and Neonatal Complications of Water-Birth Compared with Conventional Delivery. The Iranian Journal of Obstetrics, Gynecology and Infertility. 2013; 16(70):9-15.
- [Background] Nikodem VC. The effects of water birth: a randomised controlled trail. Thesis: Rand Afrikaans University, South Africa
- [Background] Alderdice F, Renfrew M, Marchant S, Ashurst H, Hughes P, Berridge G, Garcia J. Labour and birth in water in England and Wales. BMJ. 1995 Apr 1;310(6983):837. doi: 10.1136/bmj.310.6983.837. No abstract available. PMID 7711622
- [Background] Bovbjerg ML, Cheyney M, Everson C. Maternal and Newborn Outcomes Following Waterbirth: The Midwives Alliance of North America Statistics Project, 2004 to 2009 Cohort. J Midwifery Womens Health. 2016 Jan-Feb;61(1):11-20. doi: 10.1111/jmwh.12394. Epub 2016 Jan 20. PMID 26789485
- [Background] Burns EE, Boulton MG, Cluett E, Cornelius VR, Smith LA. Characteristics, interventions, and outcomes of women who used a birthing pool: a prospective observational study. Birth. 2012 Sep;39(3):192-202. doi: 10.1111/j.1523-536X.2012.00548.x. Epub 2012 Jul 3. PMID 23281901
- [Background] Demirel G, Moraloglu O, Celik IH, Erdeve O, Mollamahmutoglu L, Oguz SS, Uras N, Dilmen U. The effects of water birth on neonatal outcomes: a five-year result of a referral tertiary centre. Eur Rev Med Pharmacol Sci. 2013 May;17(10):1395-8. PMID 23740455
- [Background] Geissbühler V, Eberhard, J. Waterbirths: A Comparative Study-A Prospective Study on More than 2,000 Waterbirths. Obstetrical & gynecological survey, 2001. 56(5): 260-262.
- [Background] Zanetti-Dallenbach R, Lapaire O, Maertens A, Holzgreve W, Hosli I. Water birth, more than a trendy alternative: a prospective, observational study. Arch Gynecol Obstet. 2006 Oct;274(6):355-65. doi: 10.1007/s00404-006-0208-1. Epub 2006 Jul 26. PMID 16868755
- [Background] Taylor H, Kleine I, Bewley S, Loucaides E, Sutcliffe A. Neonatal outcomes of waterbirth: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2016 Jul;101(4):F357-65. doi: 10.1136/archdischild-2015-309600. Epub 2016 Apr 28. PMID 27127204
- [Background] Vanderlaan J, Hall PJ, Lewitt M. Neonatal outcomes with water birth: A systematic review and meta-analysis. Midwifery. 2018 Apr;59:27-38. doi: 10.1016/j.midw.2017.12.023. Epub 2017 Dec 26. No abstract available. PMID 29353689
- [Background] Gilbert RE, Tookey PA. Perinatal mortality and morbidity among babies delivered in water: surveillance study and postal survey. BMJ. 1999 Aug 21;319(7208):483-7. doi: 10.1136/bmj.319.7208.483. PMID 10454400
- [Background] Davies R, Davis D, Pearce M, Wong N. The effect of waterbirth on neonatal mortality and morbidity: a systematic review and meta-analysis. JBI Database System Rev Implement Rep. 2015 Oct;13(10):180-231. doi: 10.11124/jbisrir-2015-2105. PMID 26571292
- [Background] Dekker R, The Evidence on: Waterbirth, in Evidence Based Birth. 2018. https://evidencebasedbirth.com/waterbirth/
- [Background] Bodner K, Bodner-Adler B, Wierrani F, Mayerhofer K, Fousek C, Niedermayr A, Grunberger W. Effects of water birth on maternal and neonatal outcomes. Wien Klin Wochenschr. 2002 Jun 14;114(10-11):391-5. PMID 12708093
- [Background] Fehervary P, Lauinger-Lorsch E, Hof H, Melchert F, Bauer L, Zieger W. Water birth: microbiological colonisation of the newborn, neonatal and maternal infection rate in comparison to conventional bed deliveries. Arch Gynecol Obstet. 2004 Jul;270(1):6-9. doi: 10.1007/s00404-002-0467-4. Epub 2003 Sep 3. PMID 12955529
- [Background] Fleming SE, Donovan-Batson C, Burduli E, Barbosa-Leiker C, Hollins Martin CJ, Martin CR. Birth Satisfaction Scale/Birth Satisfaction Scale-Revised (BSS/BSS-R): A large scale United States planned home birth and birth centre survey. Midwifery. 2016 Oct;41:9-15. doi: 10.1016/j.midw.2016.07.008. Epub 2016 Jul 7. PMID 27494569
- [Background] A Model Practice Template for Hydrotherapy in Labor and Birth. J Midwifery Womens Health. 2017 Jan;62(1):120-126. doi: 10.1111/jmwh.12587. Epub 2016 Nov 24. No abstract available. PMID 27883366
- [Background] Barbosa-Leiker C, Fleming S, Hollins Martin CJ, Martin CR. Psychometric properties of the Birth Satisfaction Scale-Revised (BSS-R) for US mothers. Journal of Reproductive and Infant Psychology. 2015; 33(5):504-11.
- [Background] Hollins Martin CJ, Martin CR. Development and psychometric properties of the Birth Satisfaction Scale-Revised (BSS-R). Midwifery. 2014 Jun;30(6):610-9. doi: 10.1016/j.midw.2013.10.006. Epub 2013 Oct 24. PMID 24252712
- [Background] Fetal Heart Monitoring. J Obstet Gynecol Neonatal Nurs. 2015 Sep-Oct;44(5):683-6. doi: 10.1111/1552-6909.12743. Epub 2015 Jul 15. No abstract available. PMID 26183597
- [Background] Karimi, Laleh. Personal correspondence. (August 2019).